CLINICAL TRIAL: NCT02442622
Title: Effectiveness of Astym Treatment For de Quervain's Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-01059
Record Dates: First submitted 2015-05-08; First posted 2015-05-13 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: de Quervain's Disease
Keywords: de Quervain's disease; de Quervain's tenosynovitis.; ASTYM; de Quervain's treatment
MeSH Terms: conditions — De Quervain Disease | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Occupational therapy (Active Comparator): Traditional therapy for de Quervain's Tenosynovitis
  Interventions: Other: Occupational therapy
- Occupational therapy with ASTYM (Experimental): Traditional therapy for de Quervain's Tenosynovitis plus ASTYM
  Interventions: Device: Occupational therapy with ASTYM

INTERVENTIONS:
Other: Occupational therapy — Occupational therapy for de Quervain's Tenosynovitis
  Arms: Occupational therapy
Device: Occupational therapy with ASTYM — Occupational therapy for de Quervain's Tenosynovitis plus ASTYM
  Arms: Occupational therapy with ASTYM

SUMMARY:
To determine if the addition of Astym treatment to traditional therapy produces a more positive outcome then traditional therapy alone for the treatment of de Quervain's tenosynvitis. Two groups will be examined with one group receiving traditional therapy and the other group receiving traditional therapy in addition to Astym treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

i. Positive Finkelstein's test: The client will report pain over the first compartment of the extensor retinaculum when the thumb is tucked in the hand and deviated ulnarly.

ii. Persistent symptoms for >3 wks which have not resolved after an additional 3 weeks of splinting

iii. A diagnosis by a physician of "de Quervain's", "fist compartment tenosynovitis", or "radial styloid tenosynovitis"

iv. Patients must agree and comply to a predetermined splinting regimen

Exclusion Criteria:

i. History of cortical steroid injection to affected wrist and/or thumb

ii. History of previous wrist trauma to affected limb

iii. Comorbidity such as carpal tunnel syndrome (CTS), radial tunnel syndrome, osteoarthritis, rheumatoid arthritis, auto-immune disease or inflammatory conditions, lateral epicondylitis or tendinopathies

iv. Clotting deficits

v. Positive Cozen's sign which would indicate intersection syndrome

vi. Post-partum mothers <6 months and pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen VanLew, PhD, OTR/L, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, Center for Musculoskeletal Care, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM
Started | 15 | 17
Completed | 12 | 16
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.85 (12.57) | 42.94 (14.28) | 43.40 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 15 | 12 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale for Pain
Description: This scale is a single point scale from 0-10. The participant picks one number to represent their pain, where 0 represents no pain and 10 represents worst pain imaginable.
Time Frame: 4.5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM
Number analyzed (Participants) | 12 | 16
score on a scale | 3.2 (2.5) | 2.1 (2.7)

2. Secondary Outcome: Sequential Occupational Dexterity Assessment (SODA) Score
Description: This is a test to measure dexterity and bimanual abilities in activities of daily living. It includes 12 tasks with participants being scored on their ability, difficulty and pain during the task. Scores on the individual tasks are summed, and the range of the total SODA score is 0-108. A higher score indicates a higher dexterity.
Time Frame: 1.5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM
Number analyzed (Participants) | 12 | 16
score on a scale | 107.33 (5.6) | 106.75 (6.1)

3. Secondary Outcome: Quick Dash Score
Description: It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level. QuickDASH Scoring Formula = ([(sum of n responses)/n] -1)(25) where n represents the number of completed items. Higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score on both test ranges from 0 (no disability) to 100 (most severe disability).
Time Frame: 4.5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM
Number analyzed (Participants) | 12 | 16
score on a scale | 4.72 (5.60) | 10.61 (12.05)

ADVERSE EVENTS:
Time Frame: up to 4.5 months
Arm/Group | Occupational Therapy | Occupational Therapy With ASTYM
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT02442622/Prot_SAP_000.pdf